CLINICAL TRIAL: NCT05579964
Title: The Role of Dexmedetomidine as Myocardial Protector in Pediatric Cardiac Surgery Total Correction of Tetralogy of Fallot
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Cardiovascular Center Harapan Kita Hospital Indonesia (Other)
Responsible Party: Principal Investigator, Dian Kesumarini, MD, Principal Investigator, National Cardiovascular Center Harapan Kita Hospital Indonesia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LB.02.01/Vll/011/KEP011/2022; LB.02.01/Vll/011/KEP011/2022 (Other: National Cardiovascular Center Harapan Kita Hospital Indonesia)
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Congenital Heart Disease in Children; Cardiopulmonary Bypass; Tetralogy of Fallot
Keywords: Dexmedetomidine; Myocardial Protection; Tetralogy of Fallot; Total Correction; Double Blind Randomized Controlled Trial; Cardiopulmonary Bypass
MeSH Terms: conditions — Tetralogy of Fallot | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DEX Group (Experimental): Priming Dexmedetomidine 0.5 mcg/kg, Infusion Dexmedetomidine 0.25 mcg/kg/hour
  Interventions: Drug: Dexmedetomidine Hcl 100 Mcg/mL Inj
- Control Group (Placebo Comparator): NaCl 0.9% with adjusted amount and rate same as the DEX group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine Hcl 100 Mcg/mL Inj — Priming dose of 0.5 mcg/kg in a 5 ml syringe mixed in priming fluid and 0.25 mcg/kg/hour DEX infusion diluted in 0.9% NaCl 20 ml in a 20 ml syringe administered to the CPB reservoir with an infusion rate of 10 ml/hour
  Other Names: Precedex; Kabimidine
  Arms: DEX Group
Drug: Placebo — Priming dose of NaCl 0.9% in a 5 ml syringe mixed in priming fluid and NaCl 0.9% 20 ml in a 20 ml syringe administered to the CPB reservoir with an infusion rate of 10 ml/hour
  Other Names: NaCl 0.9%
  Arms: Control Group

SUMMARY:
Congenital heart disease (CHD) is the most common congenital abnormality found in newborns with Tetralogy of Fallot (TOF) being the most common cyanotic CHD. Total correction of TOF was performed using a cardiopulmonary bypass (CPB) machine. However, the use of CPB has a negative effect that causes inflammation and myocardial injury. Myocardial protection in patients undergoing total correction of TOF surgery is more difficult than other cyanotic CHD due to a hypertrophic right ventricular condition. Dexmedetomidine (DEX) is a selective α-2 adrenergic, which has major effects including hypnosis, sedation, and analgesia as well as cardiovascular effects. The sedation is induced by stimulating the α-2 adrenergic receptor in the locus coeruleus (LC) in the pons cerebri. DEX also increases the level of GABA and Galanin and reduces endogenous norepinephrine. The lower level of endogenous norepinephrine decreases the afterload of the ventricles, increases cardiac output, and reduces myocardial injury as a result. Furthermore, the peripheral effects of DEX can reduce myocardial ischemia-reperfusion (MIR) by inhibiting NF-кB pathway activation and reducing the number of pro-inflammatory cytokines released. Thus, the administration of DEX can prevent myocardial necrosis and apoptosis, also reducing reperfusion injury when using CPB machines. Research related to the effectiveness of administering DEX as a myocardial protector in classic TOF patients undergoing elective total correction cardiac surgery in Indonesia is less reported. The aim of this study is to determine the effectiveness of DEX as myocardial protector in classic TOF patients undergoing elective total correction cardiac surgery.

DETAILED DESCRIPTION:
This study is a double blind randomized controlled trial to determine the effectiveness of DEX during CPB as myocardial protection between DEX group and control group. The study population is classic TOF patients who underwent elective total correction cardiac surgery. This study was approved by the research ethical committee (Institutional Review Board) of the National Cardiovascular Center Harapan Kita Jakarta (NCCHK). Before randomization, participants who are eligible based on inclusion and exclusion criterias will be given informed consent. If the guardians of the participants agree, the participants will be included in this research. Sixty-six pediatric participants with classic TOF undergoing elective total correction will be randomly divided into two groups, DEX group and control group. Dexmedetomidine HCl is provided in the form of a liquid injection (Precedex/Kabimidine 200 mcg/2 ml). For the DEX group, DEX was calculated with a priming dose of 0.5 mcg/kg in a 5 ml syringe mixed in priming fluid and 0.25 mcg/kg/hour DEX infusion diluted in 0.9% NaCl 20 ml in a 20 ml syringe administered to the CPB reservoir with an infusion rate of 10 ml/hour. For the control group, the volume of administration of 0.9% NaCl as priming and 0.9% NaCl infusion was given to the CPB machine with adjusted amount and rate same as the DEX group.

We will measure myocardial injury biomarker plasma levels (Troponin I) and cytokines proinflammatory biomarkers plasma level (IL-6) as the primary outcome of myocardial protection. Serum plasma levels of troponin I and IL-6 will be taken 4 times (T1, 5 minutes after induction as baseline level; T2,1 hour after CPB; T3, 6 hours after CPB, and T4, 24 hours after CPB). Secondary outcomes including hemodynamic profile (cardiac output, cardiac index, and systemic vascular resistance, at 5 minute before induction as baseline level, 6 hours, 24 hours, and 48 hours after CPB), serum lactate levels at 5 minutes after induction as baseline level, 1 hour, 6 hours, and 24 hours after CPB, morbidity outcomes (vasoinotropic score at 1 hour, 6 hours, and 24 hours after CPB, length of ventilator use, and length of stay in intensive care).

ELIGIBILITY:
Inclusion Criteria:

* The patient's parents or person in charge is willing to participate in the study
* Patients with classic TOF undergoing elective total correction cardiac surgery
* Aged 1 month - 18 years old

Exclusion Criteria:

* The patient experiences a change in the surgical plan from elective to immediate or emergency
* Patients with preoperative infection characterized by procalcitonin >0.5ng/mL
* Patients with impaired liver function characterized by an increase in Serum Glutamic Oxaloacetic Transaminase (SGOT)/Serum Glutamic Pyruvic Transaminase (SGPT) more than 1.5 times the upper limit of normal
* Impaired renal function characterized by creatinine > 2 mg/dL
* Patients with coagulation disorders characterized by International Normalized Ratio (INR) > 1.5

Drop-out Criteria:

* Duration of CPB and/or Aortic cross-clamp time exceeding 120 minutes
* Surgery requires more than two attempts of CPB
* Patient fails to wean from CPB
* Patient requires ECMO (Extracorporeal Membrane Oxygenator) postoperatively
* Patients with postoperative reperfusion injury characterized by pulmonary hemorrhage
* Patients with residual lesions in the form of moderate-severe pulmonary stenosis and moderate-severe pulmonary regurgitation.
* Patient dies on the operating table

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-06-10 (Actual)

PRIMARY OUTCOMES:
Serum Troponin I at baseline | 5 minutes after induction of anesthesia (T1)
  Troponin I serum concentration will be measured using ELABSCIENCE E-EL-H0649 reagent (ng/mL)
Serum Troponin I at 1 hour after cardiopulmonary bypass | 1 hour after cardiopulmonary bypass (T2)
  Troponin I serum concentration will be measured using ELABSCIENCE E-EL-H0649 reagent (ng/mL)
Serum Troponin I at 6 hours after cardiopulmonary bypass | 6 hours after cardiopulmonary bypass (T3)
  Troponin I serum concentration will be measured using ELABSCIENCE E-EL-H0649 reagent (ng/mL)
Serum Troponin I at 24 hours after cardiopulmonary bypass | 24 hours after cardiopulmonary bypass (T4)
  Troponin I serum concentration will be measured using ELABSCIENCE E-EL-H0649 reagent (ng/mL)
Serum IL-6 at baseline | 5 minutes after induction of anesthesia (T1)
  IL-6 serum concentration will measured using RnD Quantikine D6050 IL-6 reagent (pg/mL)
Serum IL-6 at 1 hour after cardiopulmonary bypass | 1 hour after cardiopulmonary bypass (T2)
  IL-6 serum concentration will measured using RnD Quantikine D6050 IL-6 reagent (pg/mL)
Serum IL-6 at 6 hours after cardiopulmonary bypass | 6 hours after cardiopulmonary bypass (T3)
  IL-6 serum concentration will measured using RnD Quantikine D6050 IL-6 reagent (pg/mL)
Serum IL-6 at 24 hours after cardiopulmonary bypass | 24 hours after cardiopulmonary bypass (T4)
  IL-6 serum concentration will measured using RnD Quantikine D6050 IL-6 reagent (pg/mL)

SECONDARY OUTCOMES:
Cardiac output | 5 minutes after induction of anesthesia (T1), 6 hours (T3), 24 hours (T4), and 48 hours (T5) after cardiopulmonary bypass
  Cardiac output will be measured using transthoracic echocardiography (L/min)
Cardiac Index | 5 minutes after induction of anesthesia (T1), 6 hours (T3), 24 hours (T4), and 48 hours (T5) after cardiopulmonary bypass
  Cardiac index will be measured using transthoracic echocardiography (L/min)
Systemic Vascular Resistance (SVR) | 5 minutes after induction of anesthesia (T1), 6 hours (T3), 24 hours (T4), and 48 hours (T5) after cardiopulmonary bypass
  SVR will be measured using transthoracic echocardiography (L/min)
Serum Lactate | 5 minutes after anesthesia induction (T1), and then 1 hour (T2), 6 hours (T3), and 24 hours (T4) after cardiopulmonary bypass
  Serum lactate will be measured using an enzymatic method with a blood gas analyzer machine (mmol/L)
VIS Score | 1 hour (T2), 6 hours (T3), 24 hours (T4) after cardiopulmonary bypass
  Vasoinotropic score will be measured using the VIS formula
Mechanical ventilation time | 3 days (or until the patient is extubated)
  Mechanical ventilation time will be measured from the moment the patient arrives at the intensive care unit until the patient is extubated
Length of stay in the intensive care unit | 7 days (or until the patient is discharge from intensive care unit)
  Length of stay in the intensive care unit will be measured from the moment the patient is admitted to the intensive care unit after the surgery until discharge from intensive care unit
Mortality | 30 days post-operative
  Mortality will be measured as long as patient is hospitalized until 30 days postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Dian Kesumarini, MD, Principal Investigator — National Cardiovascular Center Harapan Kita Hospital Indonesia
Locations (1):
- National Cardiovascular Center Harapan Kita Hospital Indonesia, Jakarta, Indonesia